CLINICAL TRIAL: NCT04689737
Title: Removal of Doravirine by Hemodialysis in HIV-Infected Patients With End-Stage Renal Disease (ESRD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Dora-HD
Record Dates: First submitted 2020-12-29; First posted 2020-12-30 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2023-08

CONDITIONS: HIV-infected Participants With ESRD Undergoing Routine Hemodialysis
Keywords: HIV; ESRD; Doravirine
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — doravirine

STUDY DESIGN:
Intervention Model Description: This is a multi-centre, single-arm, open-label, pilot study in HIV-infected participants with ESRD undergoing routine hemodialysis.
  All participants will receive doravirine 100 mg once daily during the study (5 days).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Doravirine (Pifeltro, MSD) will be added to participant's cART (100 mg once daily) for 5 days
  Interventions: Drug: Doravirine

INTERVENTIONS:
Drug: Doravirine — Participants will be told to take one tablet of doravirine (Pifeltro, MDS) once daily, with or without food, approximately at the day time that they usually finish the hemodialysis sessions. The rest of their antiretroviral regimen and concomitant medications will remain unchanged
  Other Names: Pifeltro

SUMMARY:
Doravirine is a novel non-nucleoside reverse transcriptase inhibitor that has demonstrated good efficacy, tolerability, and safety for the treatment of patients with HIV infection in phase III clinical trials. Doravirine achieved non- inferiority when compared with efavirenz- and darunavir/ritonavir-based regimens. Doravirine is mainly metabolized and eliminated by the liver, with only 6% of the drug being excreted unchanged through the urine.In a study comparing 8 subjects with severe renal disease to 8 subjects without renal impairment, the single dose exposure of doravirine was 43% higher in subjects with severe renal function impairment.However, according to prescribing information, no dosage adjustment of doravirine is required in patients with mild, moderate, or severe renal impairment. On the other hand, data on doravirine pharmacokinetics in patients with ESRD on dialysis are lacking. This may be of special interest because doravirine has a relatively low molecular weight and it is only 76% bound to proteins in plasma. These characteristics could make possible for hemodialysis to remove doravirine from plasma, potentially leading to subtherapeutic concentrations of doravirine after the dialysis sessions. On the contrary, doravirine volume of distribution is about 60 liters,15 what could limit extraction of doravirine by hemodialysis. Since data on doravirine pharmacokinetics in PLWH with ESRD on dialysis are lacking, our aim is to evaluate the effect of intermittent hemodialysis on doravirine concentrations in HIV-infected patients with ESRD

DETAILED DESCRIPTION:
Doravirine is a novel non-nucleoside reverse transcriptase inhibitor that has demonstrated good efficacy, tolerability, and safety for the treatment of patients with HIV infection in phase III clinical trials. Doravirine achieved non- inferiority when compared with efavirenz- and darunavir/ritonavir-based regimens. Doravirine is mainly metabolized and eliminated by the liver, with only 6% of the drug being excreted unchanged through the urine.In a study comparing 8 subjects with severe renal disease to 8 subjects without renal impairment, the single dose exposure of doravirine was 43% higher in subjects with severe renal function impairment.However, according to prescribing information, no dosage adjustment of doravirine is required in patients with mild, moderate, or severe renal impairment. On the other hand, data on doravirine pharmacokinetics in patients with ESRD on dialysis are lacking. This may be of special interest because doravirine has a relatively low molecular weight and it is only 76% bound to proteins in plasma. These characteristics could make possible for hemodialysis to remove doravirine from plasma, potentially leading to subtherapeutic concentrations of doravirine after the dialysis sessions. On the contrary, doravirine volume of distribution is about 60 liters,15 what could limit extraction of doravirine by hemodialysis. Since data on doravirine pharmacokinetics in PLWH with ESRD on dialysis are lacking, our aim is to evaluate the effect of intermittent hemodialysis on doravirine concentrations in HIV-infected patients with ESRD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females* aging ≥ 18 years.
2. Documented HIV infection).
3. Stable antiretroviral treatment for at least 2 weeks prior to enrolment.
4. Optimal adherence to antiretroviral treatment, defined as less than 2 missed doses within the previousweek.
5. End-stage renal disease in renal replacement therapy with periodic hemodialysis.
6. Agree with the study procedures and signature of the informed consent. *Women of childbearing potential must have a negative pregnancy test prior to randomization into the study and commitment to useat least one of these birth control methods: male or female condom with or without spermicide, cap, diaphragm or sponge with orwithout spermicide, intrauterine device, bilateral tubal occlusion, vasectomized partner, sexual abstinence during the study. Condomuse is considered as an additional method of contraception only and cannot be the only method of contraception used as not beenconsidered an effective method by the Clinical Trial Facilitation Group (CTFG) guidelines.

Based on ICH, M3 (R2) 2009 a woman is considered of childbearing potential: fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include tubal ligation, hysterectomy, bilateral oophorectomy.

Exclusion Criteria:

1. Evidence or clinical suspicion that the patient will not be able to comply with the study protocol.
2. Hypersensitivity to doravirine
3. Concomitant therapy within the previous 4 weeks with any of the following drugs:

   * Anticonvulsants: carbamazepine, oxcarbazepine, phenobarbital, phenytoin
   * Androgen receptor inhibitor: enzalutamide
   * Antimycobacterials: rifampin, rifapentine
   * Cytotoxic agent: mitotane
   * St. John's wort (Hypericum perforatum)
4. Females who are pregnant or breastfeeding.
5. ALT and/ or AST ≥ 4 times the upper limit of normal (ULN) at screening.
6. Hemoglobin < 7,5 g/dL at screening.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Universitario Bellvitge Hospital, L'Hospitalet de Llobregat, Barcelona
  - Valle Hebron Hospital, Barcelona

REFERENCES:
- [Derived] Molto J, Graterol F, Curran A, Ramos N, Imaz A, Sandoval D, Perez F, Bailon L, Khoo S, Else L, Paredes R. Removal of doravirine by haemodialysis in people living with HIV with end-stage renal disease. J Antimicrob Chemother. 2022 Jun 29;77(7):1989-1991. doi: 10.1093/jac/dkac126. PMID 35425985

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Group
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentatge of Doravirine Dialysis Extraction Ratio (ER)
Description: The haemodialysis extraction ratio (ER) for doravirine was calculated as: ER(%) = ((Cin - Cout)/ Cin) × 100 where Cin is the pre-dialyser doravirine concentration (i.e. blood entering the dialyser) and Cout is the post-dialyser doravirine concentration (i.e. blood leaving the dialyser). Post-dialyser doravirine concentrations (Cout) were corrected for haemoconcentration by a factor F based on total protein (TP) concentration pre- and post-dialyser: F = TPin / TPout.
Time Frame: At day 6
Measure: Median (Full Range); unit: percentage of doravirine dialysis ER
Arm/Group | Experimental Group
Number analyzed (Participants) | 8
percentage of doravirine dialysis ER | 34.3 [25.8 to 41.4]

2. Secondary Outcome: Percentage of Participants Developing Related Adverse Events Grade 3-4 Related to Doravirine
Description: Percentage of participants developing related adverse events grade 3 or grade 4 related to doravirine. Defining Grade 3 (severe) as symptoms causing inability to perform usual social and functional activities and Grade 4 (potentially life-threatening)as Symptoms causing inability to perform basic self-care functions or Medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death.
Time Frame: Baseline to day 20
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group
Number analyzed (Participants) | 8
Participants | 2

3. Secondary Outcome: Doravirine Concentration (mg/dl)
Description: Doravirine Concentration (mg/dl) in plasma at the end of the haemodialysis session.
Time Frame: At day 6
Measure: Median (Full Range); unit: mg/dl
Arm/Group | Experimental Group
Number analyzed (Participants) | 8
mg/dl | 785 [101 to 1851]

ADVERSE EVENTS:
Time Frame: Day 1 to Day 20
Arm/Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=8)
IQ-RCFI EM Hospitalization for Fibula Fracture (Surgical and medical procedures) | 1 (1) — Hospitalization for a IQ-RCFI EM due to Fibula Fracture
Cardiac insufficiency (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=8)
Headache (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT04689737/Prot_SAP_000.pdf